CLINICAL TRIAL: NCT06824883
Title: A Single-arm, Phase 2 Study of Sintilimab, Pegaspargase Combined with Gemcitabine and Oxaliplatin (P-P-GEMOX) Regimen for Newly Diagnosed Extranodal NK/T-Cell Lymphoma
Brief Title: Sintilimab, Pegaspargase Plus GemOx for Untreated Extranodal NK/T-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NHL-019
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Extranodal NK/T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- P-P-GemOx arm (Experimental): Sintilimab, pegaspargase combined with gemcitabine and oxaliplatin (P-P-GEMOX) regimen
  Interventions: Drug: Immunochemotherapy

INTERVENTIONS:
Drug: Immunochemotherapy — P-P-GemOx regimen Sintilimab 200mg iv D1; Pegaspargase 3750U im D1; GemOx regimen: Gemcitabine 1000mg/m2 iv D1, Oxaliplatin 100mg/m2 iv D1 This regimen is administered every 3 weeks.
  For patients with stage I-II (localized) disease:
  A sandwich approach incorporating radiotherapy is employed. Patients initially receive 2 cycles of the P-P-GemOx regimen. If the interim evaluation demonstrates a complete response (CR) or partial response (PR), patients will proceed to intensity-modulated radiotherapy (IMRT). Following radiotherapy, an additional 2 cycles of the P-P-GemOx regimen are administered.
  For patients with stage III-IV (advanced) disease. Patients are planned to receive 6 cycles of the P-P-GemOx regimen. For those achieving CR or PR following 6 cycles of immunochemotherapy, subsequent treatment options include autologous hematopoietic stem cell transplantation (auto-HSCT) or PD-1 monoclonal antibody maintenance therapy, determined based on age and overall physical condition.

SUMMARY:
This is a single-arm phase 2 study designed to evaluate the safety and efficacy of sintilimab, pegaspargase combined with gemcitabine and oxaliplatin (P-P-GEMOX regimen) as first-line treatment for patients with ENKTL. The primary endpoint is the complete response rate (CRR) in the intention-to-treat population.The secondary endpoints were overall response rate (ORR), progression-free survival (PFS), overall survival (OS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of extranodal NK/T-cell lymphoma (ENKTL) by the study center.
* Age between 18 and 75 years.
* At least one of the following risk factors: Age ≥ 60 years; Presence of B symptoms; ECOG performance status ≥ 2; Elevated lactate dehydrogenase (LDH); Baseline EBV-DNA > 500 copies/mL.
* ECOG performance status of 0 to 3.
* Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L (≥ 1.0 × 10⁹/L in cases with bone marrow involvement); Platelet count (PLT) ≥ 80 × 10⁹/L (≥ 50 × 10⁹/L in cases with bone marrow involvement); Hemoglobin (HGB) ≥ 80 g/L.
* Adequate organ function: Alanine aminotransferase (ALT) < 3 × the upper limit of normal (ULN); Total bilirubin (TBil) < 1.5 × ULN; Serum creatinine < 1.5 × ULN; NYHA heart function class 0-2; Left ventricular ejection fraction (LVEF) > 50%.

Exclusion Criteria:

* Aggressive NK-cell leukemia.
* Central nervous system lymphoma.
* History of any of the following within 6 months: Acute myocardial infarction; Unstable angina; Congestive heart failure; Uncontrolled symptomatic arrhythmia; Complete left bundle branch block; Second- or third-degree atrioventricular block; Long QT syndrome or corrected QT interval (QTc) > 480 ms.
* Uncontrolled active infection.
* Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | Responses were evaluated after 3 cycles of induction and 1 month after the completion of study therapy (each cycle is 21 days)
  Treatment responses were assessed according to the 2014 Lugano classification criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of enrollment until documented disease progression or death of any reason (up to 3 years).
  Progression-free survival was defined as the time from the date of enrollment until the date of the first documented day of disease progression or relapse, or death from any cause, whichever occurred first.
Overall survival | From date of enrollment until documented death of any reason (up to 3 years).
  Overall survival was defined as the time from the date of enrollment to the date of death from any cause.
Overall response rate | Responses were evaluated after 3 cycles of induction and 1 month after the completion of study therapy (each cycle is 21 days).
  The ORR was defined as the proportion of patients with CR or PR.
Adverse event | From enrollment till 28 days post the last induction cycle.
  Graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No